CLINICAL TRIAL: NCT05381311
Title: Prospective Evaluation of Patient Preferences for Outcomes of Hormonal Agents and Chemotherapy in Combination With Androgen Deprivation Therapy
Brief Title: Survey Based Discrete Choice Experiment Study in Prostate Cancer (DECIDER) Study
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 9785-MA-3277
Record Dates: First submitted 2022-05-11; First posted 2022-05-19 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer; Metastatic Hormone-sensitive Prostate Cancer
Keywords: prostate cancer; metastatic hormone-sensitive prostate cancer; observational
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to quantify and publish participants' relative preferences for outcomes of chemotherapy and novel oral hormonal agents when added to androgen deprivation therapy (ADT) for participants with locally-advanced and metastatic hormone-sensitive prostate cancer (mHSPC). This study will also quantify the importance of administration factors related to convenience relative to treatment outcomes.

DETAILED DESCRIPTION:
The study will develop and administer a discrete-choice experiment (DCE) to quantify tradeoff preferences of participants with mHSPC and locally-advanced prostate cancer in various countries. Data/surveys are being collected in: United States, Canada, UK, France, Spain, Japan, China and South Korea.

ELIGIBILITY:
Inclusion Criteria:

For interviews (attribute prioritization and pretest interviews)

* Diagnosis of mHSPC with or without previous experience with ADT
* Able to read and understand the survey language
* Able to provide informed consent For online survey
* Diagnosis of mHSPC or locally-advanced prostate cancer with or without previous experience with ADT
* Able to read and understand the survey language
* Able to provide informed consent

Exclusion Criteria:

Not applicable

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with mHSPC or locally-advanced prostate cancer with or without previous experience with ADT.
Sampling Method: Non-Probability Sample
Enrollment: 1020 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2022-12-11 (Actual)

PRIMARY OUTCOMES:
Log-odds (preference weights) by participant cancer type and country | 1 day (once through survey)
  Log-odds indicate participants' relative preferences for treatments with each attribute level in the study, all else equal.

SECONDARY OUTCOMES:
Relative importance weights by participant type and country | 1 day (once through survey)
  These weights indicate the overall influence of each study attribute on choice.

CONTACTS AND LOCATIONS:
Overall Officials: Astellas Pharma Global Development, Inc., Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.